CLINICAL TRIAL: NCT03151564
Title: Lesion Detection Assessment in the Liver: Standard vs Low Radiation Dose Using Varied Post-Processing Techniques
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016-1135; NCI-2018-01272 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: Diseases of Liver; Colon Carcinoma; Colorectal Carcinoma; Liver Metastases
Keywords: Diseases of liver; Colon carcinoma; Colorectal carcinoma; Liver metastases; Computed tomography; CT; Reduced radiation doses; Deep Learning Image Reconstructions; DLIR
MeSH Terms: conditions — Digestive System Diseases; Colonic Neoplasms; Colorectal Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computed Tomography Scan - 50% Dose Reduction (Experimental): Participants undergo routine standard of care CT examination for colon carcinoma restaging, then have an additional scan of the liver at 50% dose reduction.
  Interventions: Diagnostic Test: Computed Tomography Scan - 50% Dose Reduction
- Computed tomography Scan - 70% Dose Reduction (Experimental): Participants undergo routine standard of care CT examination for colon carcinoma restaging, then have an additional scan of the liver at 70% dose reduction.
  Interventions: Diagnostic Test: Computed Tomography Scan - 70% Dose Reduction
- Deep Learning Image Reconstruction (DLIR) (Experimental): DLIR is available in both single (SE) and dual/multi energy (DE) CT scanning modes. DLIR SECT and DLIR DECT reconstructions have yet to be compared.
  Interventions: Diagnostic Test: Deep Learning Image Reconstruction (DLIR)

INTERVENTIONS:
Diagnostic Test: Computed Tomography Scan - 50% Dose Reduction — Participants undergo routine standard of care CT examination for colon carcinoma restaging, then have an additional scan of the liver at 50% dose reduction.
  Other Names: CT scan
  Arms: Computed Tomography Scan - 50% Dose Reduction
Diagnostic Test: Computed Tomography Scan - 70% Dose Reduction — Participants undergo routine standard of care CT examination for colon carcinoma restaging, then have an additional scan of the liver at 70% dose reduction.
  Other Names: CT scan
  Arms: Computed tomography Scan - 70% Dose Reduction
Diagnostic Test: Deep Learning Image Reconstruction (DLIR) — Participants to receive standard-of-care imaging without the artificial intelligence software and imaging technique.
  Arms: Deep Learning Image Reconstruction (DLIR)

SUMMARY:
To compare 2 different image creation/processing techniques during a standard CT scan in order to "see" problems in the liver and learn which method provides better image quality. The techniques use new artificial intelligence software to decrease image noise, which helps the radiologist to evaluate.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate whether post-processing software Adaptive Statistical Iterative Reconstruction (ASIR), ASIR-V, Veo 3.0 (GE version of Model-based Iterative Reconstruction (MBIR), and Deep Learning Image Reconstruction (DLIR) is able to preserve lesion detection in the liver and other measures of image quality at reduced radiation doses for computed tomography (CT).

Secondary Objectives:

Assessment of whether post-processing software enhances lesion detection in the liver and other measures of image quality at standard and reduced radiation doses.

Assessment of whether DLIR and GSI DLIR reconstructions perform differently, both in terms of accuracy and image quality metrics such as noise reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be >/= 18 years of age and </=90 years of age
2. Men and non-pregnant women
3. Pathology proven diagnosis of colon or colorectal carcinoma
4. Liver metastases on most recent CT examination
5. Standard of care CT abdomen examination planned WITH IV contrast

Exclusion Criteria:

1. Patients cannot give informed consent
2. Patients cannot undergo CT examination

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Metastasis Detection Accuracy | 1 day
  Primary endpoint is metastasis detection accuracy status of each patient, where the standard of care scan reviewed by ''truth readers'' (independent to the blinded radiologists) serve as the gold standard. If any lesion of a patient is diagnosed as metastasis by "truth readers" or blinded readers' consensus, that patient will be considered true positive and diagnosis positive, respectively. The expected accuracy of standard CT is 95%, and a low dose CT detection be considered non-inferior if its accuracy is 85% or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Corey T. Jensen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jensen CT, Gupta S, Saleh MM, Liu X, Wong VK, Salem U, Qiao W, Samei E, Wagner-Bartak NA. Reduced-Dose Deep Learning Reconstruction for Abdominal CT of Liver Metastases. Radiology. 2022 Apr;303(1):90-98. doi: 10.1148/radiol.211838. Epub 2022 Jan 11. PMID 35014900
- [Derived] Jensen CT, Wagner-Bartak NA, Vu LN, Liu X, Raval B, Martinez D, Wei W, Cheng Y, Samei E, Gupta S. Detection of Colorectal Hepatic Metastases Is Superior at Standard Radiation Dose CT versus Reduced Dose CT. Radiology. 2019 Feb;290(2):400-409. doi: 10.1148/radiol.2018181657. Epub 2018 Nov 27. PMID 30480489
- See also: MD Anderson Cancer Center — http://www.mdanderson.org